CLINICAL TRIAL: NCT00732732
Title: A Controlled Trail of Plantain Powder (Green Banana) in Infantile Diarrhea.
Brief Title: A Controlled Trial of Plantain Powder in Infantile Diarrhea
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Closed by US IRB due to lack of an adequate system for continuing review by the Indian IRB. No subjects enrolled in US.
Sponsor: Augusta University (Other)
Collaborators: NRS Medical College, Kolkata, West Bengal, India (Unknown); School of Tropical Medicine, Kolkata, West Bengal, India (Other)
Responsible Party: Sudipta Misra MD, Professor of Pediatrics, Medical College of Georgia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HAC 08-01-165
Record Dates: First submitted 2008-08-08; First posted 2008-08-12 (Estimated); Last update posted 2011-08-08 (Estimated); Status verified 2011-08

CONDITIONS: Diarrhea, Infantile
Keywords: diarrhea; Plantain; Green banana; Infants; Children
MeSH Terms: conditions — Diarrhea, Infantile; Diarrhea | interventions — microcrystalline cellulose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Green banana (Experimental): Subjects receiving green banana powder.
  Interventions: Dietary Supplement: Green banana powder
- Placebo (Placebo Comparator): Microcrystalline cellulose given as placebo
  Interventions: Other: Microcrystalline cellulose

INTERVENTIONS:
Dietary Supplement: Green banana powder — Green banana in powder form, 10 grams/ day for children below 10 kg, 20 grams for those weighing 10 Kg or more. Protocol Modified on Aug 5th 2009 to give 20 grams irrespective of age.
  Arms: Green banana
Other: Microcrystalline cellulose — Microcrystalline cellulose 10 gm/ day for subjects below 10 kg in weight, 20 gms/ day for those weighing 10 Kg or more
  Arms: Placebo

SUMMARY:
Green banana has been traditionally used in diarrheal and other diseases. Recent studies have shown that green banana is beneficial in children with diarrhea.

The purpose of this study is to try green banana in a portable, storable and dosable form in infants with diarrhea.

Infants with diarrhea and meeting the inclusion criteria will receive either green banana powder or placebo (microcrystalline cellulose). Their response will be monitored for 10 days. The subjects, parents and researchers conducting the study will not know whether banana powder or placebo is being given to that particular subject (double blind randomized study).

Two hundred patients will be enrolled in 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Children between the ages of 5 months and 2 years of age admitted in the inpatient pediatric ward of Bhatpara Sub divisional Hospital.
2. Infants with more than 3 stools/day which is more frequent than the usual bowel habit of the study subject
3. The consistency of the stool is such that it takes the shape of the container into which it is put in.
4. Duration of symptoms should be less than 14 days.

   -

Exclusion Criteria:

1. Children with bloody diarrhea
2. Children with lethargy, fever or other signs of septicemia
3. Children with shock.
4. Children unable to take medications orally.
5. Children with impaired consciousness.
6. Children whose parents refuse permission to be included in the study.
7. Children who are not usual residents of the area and will not be available for follow up.
8. Children with chronic illnesses such as congenital heart disease, renal failure, chronic liver disease, chronic lung disease, inflammatory bowel disease, immune deficiency etc.

   -

Ages: 5 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2008-09; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Frequency of stools per day. | Daily for 10 days

SECONDARY OUTCOMES:
Change in the consistency of stool. | Daily for 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Tapas K Sabui, MD, Principal Investigator — NRS Medical College, Kolkata.
Locations (1):
- Bhatpara Subdivisional Hospital, Bhātpāra, West Bengal, India

REFERENCES:
- [Result] Rabbani GH, Teka T, Saha SK, Zaman B, Majid N, Khatun M, Wahed MA, Fuchs GJ. Green banana and pectin improve small intestinal permeability and reduce fluid loss in Bangladeshi children with persistent diarrhea. Dig Dis Sci. 2004 Mar;49(3):475-84. doi: 10.1023/b:ddas.0000020507.25910.cf. PMID 15139502
- [Result] Rabbani GH, Teka T, Zaman B, Majid N, Khatun M, Fuchs GJ. Clinical studies in persistent diarrhea: dietary management with green banana or pectin in Bangladeshi children. Gastroenterology. 2001 Sep;121(3):554-60. doi: 10.1053/gast.2001.27178. PMID 11522739